CLINICAL TRIAL: NCT00375505
Title: Zoledronic Acid in the Prevention of Cancer Therapy Induced Bone Loss
Brief Title: The Safety and Efficacy of Zoledronic Acid in the Prevention of Cancer Therapy Induced Bone Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZOL446GDE21
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Premenopausal; Bone mineral density; Cancer therapy induced bone loss; zoledronic acid
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Zometa (Experimental): Zoledronic acid 4mg as a 15-minute infusion every 3 months for a treatment period of 24 months (total of 8 infusions).
  Interventions: Drug: Zoledronic acid
- Placebo (Placebo Comparator): Placebo as a 15-minute infusion every 3 months for a treatment period of 24 months (total of 8 infusions).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zoledronic acid
  Other Names: ZOL446, zoledronic acid, Zometa
  Arms: Zometa
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study examines the safety and efficacy of zoledronic acid 4 mg., given every 3 months over 24 months (infusion at month 0, 3, 6, 9, 12, 15, 18 and 21) in improving bone mineral density in premenopausal women with hormone receptor negative breast cancer and adjuvant chemotherapeutic treatment

ELIGIBILITY:
Inclusion Criteria:

* Female patients with histologically confirmed incident invasive breast cancer (T1-4) with positive hormone receptor status (ER and/or PgR positive) and no evidence of regional lymph node metastasis (N0) or distant metastasis (M0)
* Patient has undergone complete primary tumor resection and axillary lymph node dissection less than 90 days before start of study drug treatment.
* Patient is premenopausal at diagnosis of breast cancer (spontaneous and regular menses with premenopausal estradiol levels (>10 ng/dL)
* Patient receives adjuvant standard chemoendocrine or endocrine therapy
* Bone density at study entry > -2.5 T-Score

Exclusion Criteria:

* History of treatment or disease affecting bone metabolism (e.g., Paget's disease, primary hyperparathyroidism), prior treatment with bisphosphonates or treatments for osteoporosis in addition to calcium and vitamin D
* Abnormal renal function
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures, recent (within 6 weeks) or planned dental or jaw surgery (e.g. extraction, implants)
* Pregnancy or lactation
* Women of childbearing potential not applying a medically recognized form of contraception (i.e., oral contraceptives or implants, IUD, vaginal diaphragm or sponge, or condom with spermicide)

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (1):
- Novartis Investigative Site, Marburg, Germany

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Zometa
Started | 36 | 34
Completed | 35 | 32
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Zometa | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (6.3) | 43.2 (6.0) | 43.0 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants] — All participants were females
  Participants
    Female | 36 | 34 | 70
    Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Mineral Density (BMD) Measured by Dual (Energy) X-ray Absorptiometry (DXA) at Lumbar Spine (L2-L4) From Baseline to Month 24
Description: Bone mineral density (BMD) by DXA at lumbar spine (L2-L4); DXA assessments of the BMD at dual hips. (BMD). Two X-ray beams with different energy levels are aimed at the patient's bones. When soft tissue absorption is subtracted out, the BMD can be determined from the absorption of each beam by bone.
Time Frame: baseline, month 24
Population: ITT -Intent-To-Treat Population which contains all patients of the Safety Population for whom at least one post-baseline assessment of bone mineral density is available.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
Z-score | -0.075 (0.041) | 0.037 (0.042)

2. Primary Outcome: Change in Bone Mineral Density (BMD) at Lumbar Spine (L2-L4) From Baseline to Month 24 or Last Visit Measure by T-score
Description: Bone mineral density (BMD) at lumbar spine (L2-L4) by T-score. Your T-score is the number of units that your bone density is above or below the average. -1 and above-bone density is considered normal; Between -1 and -2.5-is a sign of osteopenia, a condition in which bone density is below normal and may lead to osteoporosis. -2.5 and below-indicates that it is likely osteoporosis.
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
T-score | -0.622 (0.346) | 0.309 (0.348)

3. Primary Outcome: Change in Bone Mineral Density (BMD) at Lumbar Spine (L2-L4) From Baseline to Month 24 or Last Visit Measure by Z-score
Description: Bone mineral density (BMD) at lumbar spine (L2-L4) measured by Z-score. If Z-score is -2 or lower, it may suggest that something other than aging is causing abnormal bone loss.
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
Z-score | -0.658 (0.355) | 0.309 (0.414)

4. Primary Outcome: Percent Change in Bone Mineral Density for L2-L4 From Baseline to Month 24 or Last Visit
Description: Bone mineral density (BMD) at lumbar spine (L2-L4) measured by using Lunar or Hologic dual-energy X-ray absorptiometry (DXA) Instruments. Measurements were done in the lumbar vertebrae (L2-L4)
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
percentage change | -6.429 (3.414) | 3.139 (3.388)

5. Secondary Outcome: Percentage Change in Bone Mineral Density for Femoral Neck (Right and Left Side) From Baseline to Month 24
Description: Bone mineral density (BMD) for femoral neck (right and left side) is measured by using Lunar or Hologic dual-energy X-ray absorptiometry (DXA) Instruments. Measurements were done on femoral neck (right and left side)
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
Percentage Change
  femoral neck (right) | -0.023 (0.033) | 0.011 (0.021)
  femoral neck (left) | -0.023 (0.035) | 0.008 (0.028)

6. Secondary Outcome: Percentage Change in Bone Mineral Density for Total Femoral Neck (Right and Left Side) From Baseline to Month 24
Description: Bone mineral density (BMD) for total femoral neck (right and left side) is measured by using Lunar or Hologic dual-energy X-ray absorptiometry (DXA) Instruments. Measurements were done on femoral neck (right and left side)
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
percentage change
  femoral neck (right) | -0.039 (0.028) | 0.013 (0.018)
  femoral neck (left) | -0.036 (0.028) | 0.014 (0.018)

7. Secondary Outcome: Change in Bone Mineral Density Os Calcis (Right and Left Side) From Baseline to Month 24 as Measured by Speed of Sound (SOS)
Description: Bone mineral density (BMD) for Os calcis (right and left side) is measured by SOS; SOS is a Quantitative ultrasonography scanning and measures bone mass and strength and assesses bone microarchitecture by detecting the transmission of high-frequency sound waves through bone.
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
m/s
  Os calcis (right) | -13.139 (23.111) | -10.853 (16.613)
  Os calcis (left) | -13.028 (19.761) | -13.485 (15.969)

8. Secondary Outcome: Change in Bone Mineral Density Os Calcis (Right and Left Side) From Baseline to Month 24 as Measured by Broadband Ultrasound Attenuation (BUA)
Description: Bone mineral density (BMD) for Os calcis (right and left side) is measured by BUA; BUA is a Quantitative ultrasonography scanning and measures bone mass and strength and assesses bone microarchitecture by detecting the transmission of high-frequency sound waves through bone.
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dB/MHz
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
dB/MHz
  Os calcis (right) | -0.306 (11.369) | 1.824 (8.997)
  Os calcis (left) | -2.417 (12.514) | 1.848 (9.628)

9. Secondary Outcome: Change in Bone Mineral Density Phalanges II, III, IV, and V From Baseline to Month 24 or Last Visit as Measured by Amplitude-dependent Speed of Sound (ADSOS)
Description: Bone mineral density (BMD) for Phalanges II, III, IV, and V is measured by ADSOS; ADSOS is a Quantitative ultrasonography scanning and measures bone mass and strength and assesses bone microarchitecture by detecting the transmission of high-frequency sound waves through bone.
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
m/s
  Phalanges II (n=35, 33) | -48.514 (50.905) | -21.485 (78.284)
  Phalanges III (n=35, 33) | -62.971 (53.760) | -19.879 (70.968)
  Phalanges IV (n=35, 33) | -49.086 (61.990) | 0.455 (93.598)
  Phalanges V (n=35, 33) | -35.000 (38.072) | 0.303 (79.985)

10. Secondary Outcome: Change in Serum CTX-carboxy-terminal Collagen Crosslinks From Baseline to Month 24
Description: CTX is a telopeptide that can be used as a biomarker in the serum to measure the rate of bone turnover. The test used to detect the CTX marker is specific to bone resorption.
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
ng/mL | 0.137 (0.164) | -0.118 (0.110)

11. Secondary Outcome: Change in Aminoterminal Propeptide on Type I Procollagen (P1NP) From Baseline to Month 24
Description: Change in Aminoterminal propeptide on type I procollagen (P1NP) from baseline to month 24. P1NP is a marker for bone formation. It is a specific indicator of type 1 collagen deposition. P1NP is increased in states of high bone turnover
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
ng/ml | 16.729 (19.346) | -21.476 (13.142)

12. Secondary Outcome: Change in Estradiol (E2) From Baseline to Month 24
Description: Change in Estradiol from baseline to month 24
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
ng/L | -119.026 (213.030) | -10.421 (134.529)

13. Secondary Outcome: Change in Follicle- Stimulating Hormone (FSH) From Baseline to Month 24
Description: Change in Follicle- Stimulating Hormone (FSH) from baseline to month 24
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mIU/ml
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
mIU/ml | -0.593 (36.851) | 0.860 (28.444)

14. Secondary Outcome: Change in Testosterone From Baseline to Month 24
Description: Change in Testosterone from baseline to month 24
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
ng/ml | 0.039 (0.110) | 0.015 (0.111)

15. Secondary Outcome: Change in Sex Hormone Binding Globulin (SHGB) From Baseline to Month 24
Description: Change in Sex Hormone binding globulin (SHGB) from baseline to month 24
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/l
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
nmol/l | 5.609 (45.614) | 12.806 (32.501)

16. Secondary Outcome: Change in Parathyroid Hormone (PTH) From Baseline to Month 24
Description: Change in Parathyroid Hormone (PTH) from baseline to month 24
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
pg/ml | 7.288 (12.838) | 4.729 (10.401)

17. Secondary Outcome: Change in Vitamine D From Baseline to Month 24
Description: Change in Vitamine D from baseline to month 24
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
ng/ml | 11.163 (9.234) | 9.638 (9.242)

18. Secondary Outcome: Change in Anti-Mueller Hormone (AMH) From Baseline to Month 24
Description: Change in anti-Mueller hormone (AMH) from baseline to month 24
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
ng/ml | -0.584 (0.962) | -0.878 (2.019)

19. Secondary Outcome: Change in Inhibin A and Inhibin B From Baseline to Month 24
Description: Change in Inhibin A and Inhibin B from baseline to month 24
Time Frame: baseline, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo | Zometa
Number analyzed (Participants) | 36 | 34
pg/ml
  Inhibin A (n=34,34) | -19.079 (29.592) | -10.209 (24.125)
  Inhibin B (n=34,34) | -28.200 (41.545) | -39.126 (43.421)

ADVERSE EVENTS:
Groups:
- Zometa: Zometa
Arm/Group | Placebo | Zometa
Serious Adverse Events (participants affected / at risk) | 3/36 | 6/34
Other Adverse Events (participants affected / at risk) | 36/36 | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | Zometa (N=34)
VERTIGO (Ear and labyrinth disorders) | 0 | 1
DENTAL CARIES (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL OEDEMA (Gastrointestinal disorders) | 1 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 1 | 0
PYREXIA (General disorders) | 1 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 1
FEBRILE INFECTION (Infections and infestations) | 0 | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
OSTEOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ATAXIA (Nervous system disorders) | 0 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1
DEPRESSION (Psychiatric disorders) | 1 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 1 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ADENOIDECTOMY (Surgical and medical procedures) | 1 | 0
HYSTERECTOMY (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | Zometa (N=34)
ANAEMIA (Blood and lymphatic system disorders) | 3 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 4 | 2
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 0
VISUAL IMPAIRMENT (Eye disorders) | 2 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 2
CONSTIPATION (Gastrointestinal disorders) | 2 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 2
NAUSEA (Gastrointestinal disorders) | 5 | 8
CHILLS (General disorders) | 1 | 7
FATIGUE (General disorders) | 1 | 2
IMPAIRED HEALING (General disorders) | 2 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 4 | 11
PYREXIA (General disorders) | 1 | 3
BRONCHITIS (Infections and infestations) | 1 | 4
CYSTITIS (Infections and infestations) | 3 | 2
GASTROENTERITIS (Infections and infestations) | 2 | 1
INFLUENZA (Infections and infestations) | 2 | 3
MASTITIS (Infections and infestations) | 2 | 0
TOOTH ABSCESS (Infections and infestations) | 1 | 2
VAGINAL INFECTION (Infections and infestations) | 2 | 0
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 2 | 0
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 0 | 2
HEPATIC ENZYME INCREASED (Investigations) | 1 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 22 | 16
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 4
BONE PAIN (Musculoskeletal and connective tissue disorders) | 12 | 11
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 2 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 5
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 2
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 | 2
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
HEADACHE (Nervous system disorders) | 3 | 6
MIGRAINE (Nervous system disorders) | 1 | 2
MOVEMENT DISORDER (Nervous system disorders) | 3 | 2
PARAESTHESIA (Nervous system disorders) | 6 | 4
DEPRESSION (Psychiatric disorders) | 1 | 5
SLEEP DISORDER (Psychiatric disorders) | 7 | 2
URGE INCONTINENCE (Renal and urinary disorders) | 1 | 2
MENOPAUSAL SYMPTOMS (Reproductive system and breast disorders) | 14 | 16
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 2
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2 | 0
HOT FLUSH (Vascular disorders) | 20 | 16
HYPERTENSION (Vascular disorders) | 3 | 2
LYMPHOEDEMA (Vascular disorders) | 19 | 11
THROMBOSIS (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety